CLINICAL TRIAL: NCT05732571
Title: Post COVID REspiratory Mechanisms and the Efficacy of a Breathing Exercise Intervention for DYsregulated Breathing (REMEDY): COVID-19
Brief Title: Post COVID-19 REspiratory Mechanisms and the Efficacy of a Breathing Exercise Intervention for DYsregulated Breathing
Acronym: REMEDY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22023; Post COVID-19 REMEDY (Other: University of Nottingham)
Record Dates: First submitted 2022-05-20; First posted 2023-02-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Respiratory Disease
MeSH Terms: conditions — COVID-19; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: A single site, pilot RCT of intervention compared to usual care
Who Masked: Outcomes Assessor
Masking Description: Randomisation will be completed in a 1:1 ratio (Intervention: Usual Care) using a sealed envelope block randomisation process.
  The study will be single blinded and controlled through the use of a distinct intervention team and an outcomes team.
  The intervention team will manage the randomisation and intervention session and planning. The outcomes team will be blinded to the intervention or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Techniques Intervention (Active Comparator): A 12 session/six week, twice a week online group-based intervention based on breathing techniques including yoga practice directed by a specialist. Each group will aim for between 3- 6 participants.
  Interventions: Other: Breathing techniques over 12 sessions / 6 weeks inc yoga
- Usual Care (No Intervention): A six week non-intervention (usual care) period will be recruited to, allowing a comparison to the intervention.

INTERVENTIONS:
Other: Breathing techniques over 12 sessions / 6 weeks inc yoga — as above
  Arms: Breathing Techniques Intervention

SUMMARY:
A pilot Study

To investigate the efficacy of a breathing intervention for improving persistent breathlessness due to dysregulated breathing following COVID-19 when compared to usual care.

DETAILED DESCRIPTION:
Pilot RCT for upto 60 subjects across 2 arms

Intervention A 12 session/six week, twice a week online group-based intervention based on breathing techniques including yoga practice directed by a specialist. Each group will aim for between 3- 6 participants.

Each online session will be circa 40-50 minutes in length. This will include an Introduction and warm up; Breathing practice including yogic breathing and a final cool down and relaxation.

Sessions will run at set times to ensure efficient use of resources but will try to accommodate different time points periods of the day when patients might be functioning best.

Comparator A six week non-intervention (usual care) period will be recruited to, allowing a comparison to the intervention.

Primary co-outcomes

Change in

* Breathlessness: Chronic Respiratory Disease Questionnaire-Dyspnoea domain (CRQ-D)
* Functional measure: 5 repetition chair to stand (5RCTS)

Secondary measures include other measures of breathlessness, function, adherence and completion (see full text for detail).

ELIGIBILITY:
Inclusion Criteria:

* Either hospitalised or non-hospitalised with confirmed COVID-19 acute infection.
* Received a comprehensive clinical respiratory assessment
* Persisting (>12 weeks) self-reported breathlessness (on CRQ-D) following COVID-19 and confirmed dysregulated breathing (Nijmegen Questionnaire score NQ >23)
* Age 18 - 80 years of age
* Ability to give informed consent
* Able to understand and speak English language

Exclusion Criteria:

* Severe mood disturbance that limits engagement with the intervention and study outcomes
* No access to online delivery and/or IT illiterate
* Significant diagnosed Myalgic Encephalitis/Fibromyalgia/Chronic Fatigue Syndrome prior to developing COVID-19
* Severe asthma or other chronic lung disease prior to COVID-19

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Breathlessness. | 7 weeks
  Chronic Respiratory Disease Questionnaire - Dyspnoea Domain Range 1-7 with lower - worse
Function | 7 weeks
  5 repetition chair to stand. Range 0-120 seconds with longer worse

SECONDARY OUTCOMES:
Dyspnoea-12 Questionnaire | 7 weeks
  SOB questionnaire. Range 0-36, Greater, worse
Nijmegen Questionnaire | 7 weeks
  Measure of dysregulated breathing. 0-64. Greater worse
Borg Scale of Breathlessness | 7 weeks
  Measure of breathlessness. Range 0-10. Greater worse
Four metre Gait speed | 7 weeks
  field test of physical performance. Range 0-60seconds. Greater worse
Modified Minnesota Physical Activity | 7 weeks
  Questionnaire. Range 0-100. Greater better.
Capnography - in some volunteers | 7 weeks
  End tidal CO2 measure in breath - at rest. Range N/A
Chalder Fatigue Score | 7 weeks
  Questionnaire. Range 0-33. Greater worse
EQ5D Quality of Life score | 7 weeks
  Questionnaire. VAS 0-100. Greater is better.
Adherence | 7 weeks
  Recorded from number of potential sessions. Range 0-12. Greater better.
Breath hold, Respiratory rate | 7 weeks
  Observational measures at rest. Breath hold - 0-45. Greater better. RR. Range 0-30. Greater worse

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bolton, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals Trust, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is pilot to generate a more formal plan